CLINICAL TRIAL: NCT00612703
Title: A Phase 1 Dose Escalation Study of ARQ 197 Administered in Combination With Erlotinib in Adult Patients With Advanced Solid Tumors
Brief Title: A Phase 1 Study of ARQ 197 in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 197-111
Record Dates: First submitted 2008-01-30; First posted 2008-02-12 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Cancer
Keywords: Cancer, oral, erlotinib, tarceva, solid tumor, advanced tumor, phase 1; Tumor
MeSH Terms: conditions — Neoplasms | interventions — ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ARQ 197 — Treatment with ARQ 197 in combination with erlotinib

SUMMARY:
To determine the safety, tolerability and recommended Phase 2 dose of ARQ 197 when administered in combination with erlotinib to patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent must be obtained and documented according to International Conference on Harmonization (ICH)- Good Clinical Practice (GCP), the local regulatory requirements, and permission to use private health information in accordance with the Health Insurance Portability and Accountability Act (HIPPA) prior to study-specific screening procedures
* A histologically or cytologically confirmed solid tumor that is advanced, metastatic, and/or inoperable following prior standard chemotherapy, and/or for which, in the opinion of the investigator, there is no alternative therapy, or for which monotherapy with erlotinib is appropriate
* ≥ 18 years of age
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST)

Exclusion Criteria:

* Anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within four weeks of first dose (patients currently on erlotinib monotherapy may be enrolled into the study without a washout)
* Major surgery within 4 weeks prior to first dose
* Central nervous system metastasis unless it has been stable for ≥ 3 months after treatment and patient has no neural symptoms
* Pregnant or breastfeeding
* Significant gastrointestinal disorder that, in the opinion of the Investigator, could interfere with the absorption of ARQ 197 and/or erlotinib (e.g. significant, uncontrolled inflammatory bowel disease or extensive small bowel resection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-02; Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability and recommended Phase 2 dose of ARQ 197 when administered in combination with erlotinib to patients with advanced solid tumors | No time frame

SECONDARY OUTCOMES:
To determine the pharmacokinetic profiles of ARQ 197 and erlotinib, when administered in combination to patients with advanced solid tumors | No time frame
To assess the preliminary anti-tumor activity of ARQ 197 when administered in combination with erlotinib to adult patients with advanced solid tumors | No time frame

CONTACTS AND LOCATIONS:
Overall Officials: Lee Rosen, MD, Principal Investigator — Premiere Oncology of Santa Monica; Richard G Just, MD, Principal Investigator — Pacific Oncology and Hematology Associates
Locations (2):
- United States (2):
  - San Diego Pacific Oncology and Hematology Associates Inc., Encinitas, California
  - Premiere Oncology, Santa Monica, California

REFERENCES:
- [Derived] Goldman JW, Laux I, Chai F, Savage RE, Ferrari D, Garmey EG, Just RG, Rosen LS. Phase 1 dose-escalation trial evaluating the combination of the selective MET (mesenchymal-epithelial transition factor) inhibitor tivantinib (ARQ 197) plus erlotinib. Cancer. 2012 Dec 1;118(23):5903-11. doi: 10.1002/cncr.27575. Epub 2012 May 17. PMID 22605616